CLINICAL TRIAL: NCT04921072
Title: Neuroplasticity in Motor Learning Under Variable and Constant Practice Conditions
Brief Title: Neuroplasticity in Motor Learning in Young Adults Under Variable and Constant Practice Conditions
Acronym: NMLPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: Czech-BioImaging (Unknown); Wroclaw University of Health and Sport Sciences (Other)
Responsible Party: Principal Investigator, Stanisław Henryk Czyż, Principal Investigator, Masaryk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FSpS SHC 1
Record Dates: First submitted 2021-06-03; First posted 2021-06-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Neuroplasticity in Motor Learning
Keywords: sensorimotor cortex activity; neuroplasticity; specificity of practice; variability of practice; practice conditions; motor learning

STUDY DESIGN:
Intervention Model Description: Fifty participants will be randomly assigned to two groups: constant and variable practice condition group (CG and VG). The pretest-posttest design will be applied.
  All participants will go through MRI scanning and EEG measurements. All participants will perform a pretest (baseline) consisting of 15 trials of SPSIC (1-3) and MRCP - motor related cortical potential, as the specific type of event related potential. The testing will start with MRCP, then SPSIC 1, then SPSIC 2, and will finish with SPSIC 3. The testing will be scheduled in blocked order. After completing the whole training program, each participant will perform a posttest analogically to the pretest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CG - Constant practice condition group (Experimental): CG will be practicing only one specific pattern of step isometric contractions (SPSIC) scheme. It means that 90 trials in all training sessions will consist only of SPSIC 1.
  Interventions: Behavioral: Constant practice conditions
- VG - Variable practice condition group (Experimental): VG will practice three SPSIC's (1-3). Each SPSIC will be practiced 30 times per session, which means that each session will consist of 90 SPSIC like CG.
  Interventions: Behavioral: Variable practice conditions

INTERVENTIONS:
Behavioral: Constant practice conditions — CG will be practicing only one specific pattern of step isometric contractions (SPSIC) scheme. It means that 90 trials in all training sessions will consist only of SPSIC 1.
  Arms: CG - Constant practice condition group
Behavioral: Variable practice conditions — VG will practice three SPSIC's (1-3). Each SPSIC will be practiced 30 times per session, which means that each session will consist of 90 SPSIC like CG.
  Arms: VG - Variable practice condition group

SUMMARY:
The project aims at providing a better understanding of motor skill acquisition and learning processes.

The primary objectives of the study are to determine how practice conditions, i.e., variable and constant practice conditions, in motor learning affect Central Nervous System. There are three objectives:

1. to determine functional changes following constant and variable practice conditions in motor learning (resting-state fMRI)
2. to determine the EEG activation and connectivity between cognitive, sensory, and motor cerebral cortex areas (central, temporal, parietal, occipital) in constant and variable practice conditions and as a function of practice time.

DETAILED DESCRIPTION:
Variable practice involving the practice of several variations of motor skill benefits learning differently than practice in constant conditions, i.e., practice that involves only one variation of a skill. The variable practice results in better retention and transfer. The performance of a skill practiced in variable conditions is more accurate and stable. In contrast, practicing only one variation of a skill better refines the recall schema. It means that the motor program (which serves as an "example" while executing a movement) is developed better. The trained variation of a skill (in constant practice), produces an advantage in performance compared to the same variation of the skill that was practiced in variable conditions (assuming that variable and constant practice had similar capacity).

This finding has an important implication for those who want to master their skills and it does not matter whether this skill refers to sport, driving, piloting, or rehabilitation. If one wants to be good at performing only one variation of a skill, one should practice in constant conditions, whereas if one wants to be good in more than one variation of skill and wants to generalize the experience to novel situations an individual should practice in variable conditions. As one can see, this implication is practical, although the mechanisms underlying this distinction and differences are unknown.

On the other hand, it is unquestioned today that learning new motor skills dynamically changes brain, i.e., brain is neuroplastic. The neuroplasticity of the brain is specifically conspicuous in the progression of motor learning. As it was reported in previous research, cortico-striatal and cortico-cerebellar systems play an important role in motor skill acquisition. However, both of these systems differ in terms of the role they play as learning progresses. Cortico-striatal system (associative/premotor brain regions) is primarily engaged in the initial phase of learning, i.e., in cognitive functioning and sensory processing. Cortico-cerebellar system (sensorimotor network) is becoming more active in the later phase of motor learning. However, none of the previous research focused on what role these systems play in learning under different conditions and how the different roles the systems may play affect structural neuroplasticity, including grey and white matter.

It may be also interesting to look at the functional neuroplasticity. A lesser degree of cognitive involvement during the execution of movements may be associated with lower activation in the sensorimotor cortex. On the other hand, increased cognitive involvement may be expected in variable conditions due to, e.g., stimulus identification or decision making. Therefore, the assumption that decreased cognitive involvement and, as a result, decreased prefrontal cortex activation in constant practice conditions sounds reasonable. Moreover, it may be hypothesized that practicing and learning in constant conditions will be characterized by lower sensorimotor cortex activation since there will be decreased control during the motor performance, which leads to more adaptive motor performance.

ELIGIBILITY:
Inclusion Criteria:

* no history of epilepsy, any known neurological disorder, no psychiatric history, were medication-free during the previous 14-days prior to participation, had not used alcohol within the previous 24-h and were not pregnant

Exclusion Criteria:

* Participants will be excluded if they were a musician or a professional typist, or had any contraindications to MRI, significant medical conditions that prevented them from performing the task, or scored less than 3 on the Mini-Cog ™ test.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional changes following constant and variable practice conditions in motor learning (resting state fMRI) | pretest - 3 and 4 weeks posttests
  Structural, diffusion, and resting-state functional scans will be acquired both prior to and after the three weeks of practicing the unimanual index finger abduction motor task. High-resolution T1-weighted (MPRAGE) and FLAIR images will be exploited to assess grey matter changes. Diffusion-weighted (DWI) data will be used for probabilistic tractography to obtain specific tracts that will be analyzed in terms of alterations in fractional anisotropy, mean, radial, and parallel diffusivity. In addition, whole-brain white matter microstructural changes will be assessed using Tract-Based Spatial Statistics (TBSS).
  Regarding resting-state fMRI data, BOLD multi-echo echo-planar imaging fMRI sequence will be applied.
SMR differences in constant and variable practice conditions in motor learning and as a function of practice time | pretest - 3 and 4 weeks posttests
  To test the sensorimotor cortex activity and coherence in constant and variable practice conditions, the sensorimotor rhythm (SMR) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stanisław H. Czyż, Ph.D., Principal Investigator — Masaryk University, Brno, Czech Republic
Locations (1):
- Masaryk University, Faculty of Sport Studies, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
All anonymized IPD will be shared using one of the many open repositories, however, how the data will be organized and how it will be presented has to be decided (given the complexity and amount of imaging data).

REFERENCES:
- [Derived] Czyz SH, Marusiak J, Klobusiakova P, Sajdlova Z, Rektorova I. Neuroplasticity in Motor Learning Under Variable and Constant Practice Conditions-Protocol of Randomized Controlled Trial. Front Hum Neurosci. 2022 Mar 17;16:773730. doi: 10.3389/fnhum.2022.773730. eCollection 2022. PMID 35370573